CLINICAL TRIAL: NCT05430737
Title: A Phase II Clinical Study of Stereotactic Radiation Therapy Based on Multiparameter Magnetic Resonance Image in Patients With High-risk Prostate Cancer
Brief Title: A Phase II Clinical Study of Stereotactic Radiation Therapy in Patients With High-risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wang Xin, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-PCa-001
Record Dates: First submitted 2022-05-26; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer; Stereotactic Body Radiotherapy; High-risk; Efficacy; Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiotherapy (Experimental): Long-term ADT of 2-3years were administered. Neoadjuvant ADT within 6 months was allowed.Then patients with high-risk prostate cancer recieve stereotactic body radiotherapy with pelvic radiation and GTV boost based on multiparameter magnetic resonance image.
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — The radiation dose to the primary tumor was 40 or 45 Gy in five fractions according to the clinical determination of the radiologist. The dose to the positive lymph nodes and the prostate and seminal vesicles was 37.5Gy in five fraction. And internal iliac, external iliac, obturator, and presacral pelvic drainage regions received 25 Gy/5f, simultaneously. The treatment was delivered every other day. The volumetric modulated arc radiotherapy (VMAT) or intensity-modulated radiotherapy (IMRT) was used to complete treatment. Image-guided radiotherapy(IGRT) was performed for every treatment.

SUMMARY:
Stereotactic body radiotherapy (SBRT) has emerged as an effective and safe treatment for low and intermediate-risk prostate cancer(PCa). However, there is no study that has investigated the effectiveness and safety of SBRT with pelvic radiation and gross target volume(GTV) boost for high-risk prostate cancer patients yet. The investigators designed a phase II clinical study of SBRT with pelvic radiation and GTV boost based on mpMRI in patients with high-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* pathologically confirmed high-risk (T3a or Gleason score ≥ 8 or a PSA > 20 ng/ml) prostate cancer
* a WHO performance status 0-1
* history of neoadjuvant androgen deprivation therapy(ADT) within 6 months before enrollment
* Patients with pelvic positive lymph node were also included in our study

Exclusion Criteria:

* distant metastasis
* history of neoadjuvant ADT over 6 months before enrollment
* history of definitive treatment for prostate cancer such as radical prostatectomy
* history of pelvic irradiation; prostate volume≥100 cm3

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
biochemical relapse-free survival | three months
  2-years biochemical relapse-free survival

SECONDARY OUTCOMES:
the incidence rate of acute toxicity | every week
  the incidence rate of toxicity in 90 days
the incidence rate of late toxicity | three months
  the incidence rate of toxicity after 90 days
patient-reported quality of life | three months
  patient-reported quality of life using European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30(EORTC QLQ C30) .The The minimum and maximum values of EORTC QLQ C30 are 0 and 100,respectively.Higher scores for functional and overall health areas of EORTC QLQ C30 indicate better functional status and quality of life, and higher scores for symptom areas indicate more symptoms or problems.
symptom score | three months
  Symptom score using the International Prostatic System Score (IPSS) .The minimum and maximum values of IPSS are 0 and 35,respectively.A higher score of IPSS means a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: xin wang, Principal Investigator — China, SiChuan West China Hospital
Locations (1):
- China, SiChuan, Chengdu, Sichuan, China